CLINICAL TRIAL: NCT02029144
Title: Dydrogesterone in Cycle Regularization in Abnormal Uterine Bleeding - Ovulation Dysfunction (AUB-O) Patients: A Prospective, Observational Study
Brief Title: Observational Study of Dydrogesterone in Cycle Regularization
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Zhang Wei, Professor, Fudan University
Other Study IDs: A14-390
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Observational Study; Dydrogesterone; Irregular Menstrual Cycle; Abnormal Uterine Bleeding
MeSH Terms: conditions — Menstruation Disturbances; Metrorrhagia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Dydrogesterone has been widely used worldwide for various gynecological and obstetric indications:

* Dydrogesterone is effective in cycle regulation treatment.
* Dydrogesterone is recognized as none interference to hypothalamus pituitary ovary (HPO) axis in the recommended dosage.
* Dydrogesterone might have non-negative effect on glucose and lipid metabolic.

DETAILED DESCRIPTION:
The current study is designed as a prospective, non-interventional, observational study. Patients with irregular cycle diagnosed as AUB-O will be prescribed dydrogesterone as per physician's clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16 years or above with menses
* Patient who is suffering from irregular menstrual cycle for at least 3 months and has been diagnosed as AUB-O (irregular cycle is defined as cycle duration < 21days or >35 days)
* Physicians have decided to prescribe dydrogesterone 10mg for cycle regulation treatment, orally taking dydrogesterone 10mg twice daily, from day16 to day 25 of each cycle, being consecutive at least 3 cycles
* Patient who is willing to sign written authorization

Exclusion Criteria:

* Hyperprolactinemia and thyroid dysfunction.
* Patient took cycle regulation treatment including oral contraceptives, sex hormone or glucocorticoid in the past 1 month
* Women with estrogen deficiency related symptom
* Patient who meets the contraindications listed in Chinese label of dydrogesterone
* Pregnant and lactating patients
* Patient who is not suitable for the study according to physician's discretion

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese women who is suffering from irregular menstrual cycle for at least 3 months and has been diagnosed as AUB-O
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
percentage of patients reporting a regular cycle (defined as cycle duration≥21 and ≤ 35 days) at the end of cycle 3 | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality, China